CLINICAL TRIAL: NCT03096548
Title: Sun Safety Ink! A Sun Safety Program for the Tattoo Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0315; R01CA206569 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-03-30 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Skin Cancer
Keywords: Skin Cancer; Tattoo
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sun Safety Ink! Program (Experimental): A program to (1) increase full-body sun comprehensive sun protection practices, (2) decrease sunburning and tanning and (3) decrease positive attitudes regarding tanning and tanning attractiveness of tattoo studio clients. The program is comprised of a video based communication strategy training presented by research staff to artists of tattoo studios.
  Interventions: Behavioral: Sun Safety Ink! Program
- Attention Control (Active Comparator): The attention control group will provide standard tattoo aftercare instructions to their clients.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Sun Safety Ink! Program — The intervention will be comprised of an online skin cancer prevention training for all tattoo artists of participating studios. The training will include skin cancer rates and risk factors, tattoo rates, recommendations for sun protection practices, a rationale for the relationship of tattoo care and sun safety, and recommended communication strategies for artists to communicate skin cancer prevention to their clients. Additional printed materials (tip-card for clients, posters) to be displayed in tattoo studios, a Sun Safety Ink! website, and social media messages for tattoo studios' Facebook and Pinterest pages will be provided.
  Arms: Sun Safety Ink! Program
Behavioral: Attention Control — Studios and artists in this attention control group will not receive the Sun Safety Ink! program. They will continue to provide standard aftercare instructions to clients. The program will be provided to them at the end of the study.
  Arms: Attention Control

SUMMARY:
Over 3.5 million cases of non-melanoma skin cancers occur annually and melanoma rates have doubled in the last 30 years, burdening the nation's health system. Klein Buendel, Inc. (KB) proposes to develop Sun Safety INK! (SSI!), a skin cancer prevention program targeted to clients of licensed tattoo studios because tattoo aftercare recommendations can include sun protection for tattoos, and studios offer an opportunity to reach younger adults who are significantly more likely to sunburn and less likely to practice sun safety. The study will assess the effectiveness of SSI! at (1) increasing full-body comprehensive sun protection practices; (2) decreasing sun burning and tanning; and, (3) decreasing positive attitudes regarding tanning and tanning attractiveness.

DETAILED DESCRIPTION:
Skin cancer prevention is a public health priority. Over 3.5 million cases of non-melanoma skin cancers (NMSC) occur annually and melanoma rates have doubled in the last 30 years, burdening the nation's health system. Increasing evidence points to the need for prevention programs to be targeted to young adults as invasive melanoma of the skin is the third most common cancer among adolescents and young adults (ages 15-39) in the U.S. Skin cancer is preventable as excess exposure to ultraviolet radiation (UVR), the primary risk factor, is modifiable and a number of public health campaigns have been developed to increase awareness about skin cancer risk and to promote sun safety. Despite these efforts, skin cancer rates continue to rise. Many adults still forget to apply sunscreen, do not pre-apply prior to sun exposure, fail to reapply, do not use clothing or wide-brimmed hats that physically block UVR and do not use shade. 4.2% of US adults engage in indoor tanning. It is well established that continued efforts are needed to promote skin cancer prevention. Concurrently, approximately, 25% of American adults have a tattoo with younger adults more likely to have tattoos than older adults. The popularity of tattoos continues to grow in the general population and particularly among members of the military. Individuals with tattoos need to take extra precaution when exposed to the sun not only to protect themselves from harmful UVR rays but also to reduce damage to their tattoos. Klein Buendel, Inc. (KB) proposes to develop and test Sun Safety INK (SSI), a skin cancer prevention program targeted to clients of licensed tattoo studios. The studios have been selected as the venue for this study because tattoo salons, at times, promote sun protection for new tattoos to keep them from fading, and offer a unique opportunity to reach younger adults who have high sunburn rates and are often less likely to practice sun protection. The studios provide a unique and compatible environment for sun safety promotion. Further, a number of successful programs have promoted health practices through similar venues such as beauty parlors and barber shops. Exploratory research with the tattoo community determined that: (1) tattoo studios were receptive to a skin cancer prevention program; (2) tattooed individuals had high rates of sunburns and low rates of sun protection but were open to receiving sun safety information and (3) a prototype SSI! program confirmed feasibility for recruitment and implementation. Based on these results, KB proposes to fully develop SSI! to include an online sun safety training for artists, a website, and additional sun safety education materials (e.g., social media). KB will work with the Alliance of Professional Tattoo Artists and the National Tattoo Association to recruit 30 licensed studios to participate in a group-randomized pair-matched pretest-posttest controlled quasi-experimental design. The primary outcomes of the study will be to evaluate the effectiveness of SSI! at: (1) increasing full-body comprehensive sun protection practices; (2) decreasing sun burning and tanning; and, (3) decreasing positive attitudes regarding tanning and tanning attractiveness.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must have received a tattoo in a licensed tattoo studio

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1820 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Sun Protection by Client (online survey) | Baseline, 1 Month Posttest, 6 Month Posttest
  Sun protection practices (sunscreen application/reapplication and Sun Protection Factor (SPF); use of lip balm, hats, protective clothing, sunglasses, shade) of tattooed and non-tattooed skin will be assessed in an online survey.
Change in Number of Sunburns | Baseline, 1 Month Posttest, 6 Month Posttest
  Participants will report number of sunburns in the past 12 months.

SECONDARY OUTCOMES:
Change in Tanning Behaviors (online survey) | Baseline, 1 Month Posttest, 6 Month Posttest
  Participants will complete an online survey that focuses on tanning frequency for both indoor and outdoor tanning.
Change in Tanning Attitudes (online survey) | Baseline, 1 Month Posttest, 6 Month Posttest
  Participants will complete an online survey that focuses on a six-item tanning image scale (1= strongly agree to 5= strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Walkosz, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Klein Buendel, Inc., Golden, Colorado

IPD SHARING:
Plan to Share IPD: No